CLINICAL TRIAL: NCT06288230
Title: Study of AAV-hSMN1 (Vesemnogene Lantuparvovec) Gene Therapy in Subjects With Progressive Spinal Muscular Atrophy
Brief Title: An Open Label Study of Gene Therapy Product (Vesemnogene Lantuparvovec) in Spinal Muscular Atrophy
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Lantu Biopharma (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: LT01-101
Record Dates: First submitted 2024-02-18; First posted 2024-03-01 (Actual); Last update posted 2025-07-22 (Actual); Status verified 2025-07

CONDITIONS: Spinal Muscular Atrophy
MeSH Terms: conditions — Muscular Atrophy, Spinal

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Stage 1: Dose A in children < 24 months of age (Experimental): Dose escalting study: Administration Dose A of Vesemnogene Lantuparvovec in children < 24 months of age
  Interventions: Biological: vesemnogene lantuparvovec
- Stage 1: Dose B in children < 24 months of age (Experimental): Dose escalting study: Administration Dose B of Vesemnogene Lantuparvovec in children < 24 months of age
  Interventions: Biological: vesemnogene lantuparvovec
- Stage 2: The selected dose in children ≥ 24 months of age (Experimental): Administration the selected dose of Vesemnogene Lantuparvovec in children ≥ 24 months of age
  Interventions: Biological: vesemnogene lantuparvovec

INTERVENTIONS:
Biological: vesemnogene lantuparvovec — Exploratory study evaluating the safety and efficacy of vesemnogene lantuparvovec in patients with SMA.
  Other Names: AAV-hSMN1

SUMMARY:
This is an interventional study to evaluate safety and efficacy of AAV-hSMN1 in spinal muscular atrophy patients.

DETAILED DESCRIPTION:
Study duration per participant is approximately 25 months including an approximately 30-day screening/baseline period, an approximately 24-month study observation period including 1 treatment day, and an approximately 24-month follow-up period. Patients will be stratified in two groups, those < 24 months of age at time of dosing and those ≥ 24 months of age at time of dosing. This study will be conducted in 2 stages:

Stage 1: dose escalting study in children <24 months of age. Stage 2: the selecetd dose from Stage 1 in children ≥ 24 months of age.

Patients will be tested at baseline and return for follow-up visits twice a week through the first month post dose, and followed by visits at months 2, 3, 6 12, 18 and 24 post infusion. Unscheduled visits may occur if the investigator determines that they are necessary.

For patients enrolled from overseas, follow-up visits with patient's own paediatrician together with remote virtual visits are allowed.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of SMA based on gene mutation analysis with bi-allelic survival motor neuron (SMN1) mutations (deletion or point mutations).
* Patients or Parent(s)/legal guardian(s) willing and able to complete the informed consent process and comply with study procedures and visit schedule.

Exclusion Criteria:

* Anti-AAV9 antibody titers >1:20 as determined by Enzyme-linked Immunosorbent Assay (ELISA) binding immunoassay.
* Active viral infection (includes HIV or serology positive for hepatitis B or C).
* Use of invasive ventilatory support (tracheotomy with positive pressure) or pulse oximetry <95% saturation.
* Concomitant illness and any drug that in the opinion of the investigator creates unnecessary risks for gene transfer.
* Clinically significant abnormal laboratory values.
* Participation in a recent SMA treatment clinical trial that in the opinion of the PI creates unnecessary risks for gene transfer.
* Patient with signs of aspiration based on a swallowing test and unwilling to use an alternative method to oral feeding.
* For children ≥ 24 months of age, contraindications for spinal tap procedure or administration of intrathecal therapy or presence of an implanted shunt for the drainage of CSF or an implanted central venous (CNS) catheter.
* For children ≥ 24 months of age, severe contractures as determined by Physical Therapist(s) at screening that interfere with either the ability to attain/demonstrate functional measures or interferes with ability to receive dosing.
* For children ≥ 24 months of age, severe scoliosis (defined as ≥ 50° curvature of spine) evident on X-ray examination.
* For children ≥ 24 months of age, previous, planned or expected scoliosis repair surgery/procedure within 1 year of dose administration.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2024-10-20 (Actual); Primary Completion 2027-10-30 (Estimated); Study Completion 2027-10-30 (Estimated)

PRIMARY OUTCOMES:
Numbers of participants with adverse events (AEs), serious adverse events (SAEs) | Baseline up to 24 months
  Participants are monitored for safety from baseline up to the end of the follow-up period.

SECONDARY OUTCOMES:
Change from baseline in developmental gross motor milestones achieved according to WHO criteria | Baseline up to 24 months
  For patients with SMA, the percentage of participants who are able to preserve ambulatory function.
Change from baseline in CHOP-INTEND in children <24 months of age | Baseline up to 24 months
  The CHOP-INTEND contains 16 items rated from 0 to 4. Total scores range from 0-64. Higher scores indicate higher levels of motor ability.
Change from baseline in Hammersmith Functional Motor Scale - Expanded (HFMSE) in children ≥ 24 months of age | Baseline up to 24 months
  The HFMSE contains 33 items rated from 0 (unable to perform) to 2 (performs without modification/adaptation/compensation). Total scores range from 0-66. Higher scores indicate higher levels of motor ability.

CONTACTS AND LOCATIONS:
Locations (1):
- Kunming Hope of Health Hospital, Kunming, Yunnan, China